CLINICAL TRIAL: NCT01294449
Title: Multicenter Automatic Defibrillator Implantation Trial With Cardiac Resynchronization Therapy Post Approval Registry
Acronym: MADIT-CRT PAR
Status: Completed | Type: Observational
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: MADIT-CRT PAR
Record Dates: First submitted 2011-02-07; First posted 2011-02-11 (Estimated); Results first posted 2014-12-04 (Estimated); Last update posted 2014-12-04 (Estimated); Status verified 2014-03

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- MADIT-CRT ICD
  Interventions: Device: MADIT-CRT ICD
- MADIT-CRT CRT-D
  Interventions: Device: MADIT-CRT CRT-D

INTERVENTIONS:
Device: MADIT-CRT ICD — Patients that were randomized to the the implantable cardioverter defibrillator (ICD) device for the study.
  Other Names: Market approved Boston Scientific implantable cardioverter defibrillators
  Groups: MADIT-CRT ICD
Device: MADIT-CRT CRT-D — Patients that were randomized to the the cardiac resynchronization therapy with defibrillation (CRT-D) device for the study.
  Other Names: Boston Scientific market approved cardiac resynchronization therapy defibrillators
  Groups: MADIT-CRT CRT-D

SUMMARY:
MADIT-CRT PAR is an FDA mandated follow-up registry for patients that participated in the MADIT-CRT IDE study examining long-term mortality.

(MADIT-CRT IDE: NCT00180271)

DETAILED DESCRIPTION:
The registry is designed to determine the long-term mortality benefit as a result of Cardiac Resynchronization Therapy with Defibrillation (CRT-D) vs. Implantable Cardioverter Defibrillator (ICD) therapy in the MADIT-CRT study patient population. The registry will collect data on patients that previously participated at MADIT-CRT sites within the US through five years of participation from their orginal enrollment in the MADIT-CRT IDE study (MADIT-CRT IDE: NCT00180271).

ELIGIBILITY:
Inclusion Criteria:

* Active patients who were enrolled in the MADIT-CRT IDE (NCT00180271)within the United States

Exclusion Criteria:

* Patients who are unable or unwilling to comply with the protocol requirements

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The registry involves only those patients that participated in the MADIT-CRT IDE study within the United States.
Sampling Method: Probability Sample
Enrollment: 394 (Actual)
Dates: Start 2011-03; Primary Completion 2013-10 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Arthur J Moss, MD, Principal Investigator — University of Rochester Heart Research Follow-up Program
Locations (1):
- University of Rochester /Strong Memorial, Rochester, New York, United States

REFERENCES:
- [Derived] Vidula H, Lee E, McNitt S, Polonsky B, Aktas M, Rosero S, Younis A, Solomon SD, Zareba W, Kutyifa V, Goldenberg I. Cardiac Resynchronization Therapy and Risk of Recurrent Hospitalizations in Patients Without Left Bundle Branch Block: The Long-Term Multicenter Automatic Defibrillator Implantation Trial With Cardiac Resynchronization Therapy. Circ Heart Fail. 2020 Jul;13(7):e006925. doi: 10.1161/CIRCHEARTFAILURE.120.006925. Epub 2020 Jul 1. PMID 32605387
- [Derived] Kutyifa V, Vermilye K, Solomon SD, McNitt S, Moss AJ, Daimee UA. Long-term outcomes of cardiac resynchronization therapy by left ventricular ejection fraction. Eur J Heart Fail. 2019 Mar;21(3):360-369. doi: 10.1002/ejhf.1357. Epub 2018 Dec 28. PMID 30592353
- [Derived] Biton Y, Kutyifa V, Cygankiewicz I, Goldenberg I, Klein H, McNitt S, Polonsky B, Ruwald AC, Ruwald MH, Moss AJ, Zareba W. Relation of QRS Duration to Clinical Benefit of Cardiac Resynchronization Therapy in Mild Heart Failure Patients Without Left Bundle Branch Block: The Multicenter Automatic Defibrillator Implantation Trial with Cardiac Resynchronization Therapy Substudy. Circ Heart Fail. 2016 Feb;9(2):e002667. doi: 10.1161/CIRCHEARTFAILURE.115.002667. PMID 26823498
- [Derived] Biton Y, Zareba W, Goldenberg I, Klein H, McNitt S, Polonsky B, Moss AJ, Kutyifa V; MADIT-CRT Executive Committee. Sex Differences in Long-Term Outcomes With Cardiac Resynchronization Therapy in Mild Heart Failure Patients With Left Bundle Branch Block. J Am Heart Assoc. 2015 Jun 29;4(7):e002013. doi: 10.1161/JAHA.115.002013. PMID 26124205
- [Derived] Daimee UA, Moss AJ, Biton Y, Solomon SD, Klein HU, McNitt S, Polonsky B, Zareba W, Goldenberg I, Kutyifa V. Long-Term Outcomes With Cardiac Resynchronization Therapy in Patients With Mild Heart Failure With Moderate Renal Dysfunction. Circ Heart Fail. 2015 Jul;8(4):725-32. doi: 10.1161/CIRCHEARTFAILURE.115.002082. Epub 2015 Jun 2. PMID 26038537
- [Derived] Goldenberg I, Kutyifa V, Klein HU, Cannom DS, Brown MW, Dan A, Daubert JP, Estes NA 3rd, Foster E, Greenberg H, Kautzner J, Klempfner R, Kuniss M, Merkely B, Pfeffer MA, Quesada A, Viskin S, McNitt S, Polonsky B, Ghanem A, Solomon SD, Wilber D, Zareba W, Moss AJ. Survival with cardiac-resynchronization therapy in mild heart failure. N Engl J Med. 2014 May 1;370(18):1694-701. doi: 10.1056/NEJMoa1401426. Epub 2014 Mar 30. PMID 24678999
- [Derived] Skali H, Dwyer EM, Goldstein R, Haigney M, Krone R, Kukin M, Lichstein E, McNitt S, Moss AJ, Pfeffer MA, Solomon SD. Prognosis and response to therapy of first inpatient and outpatient heart failure event in a heart failure clinical trial: MADIT-CRT. Eur J Heart Fail. 2014 May;16(5):560-5. doi: 10.1002/ejhf.71. Epub 2014 Feb 27. PMID 24578164
- [Derived] Campbell P, Takeuchi M, Bourgoun M, Shah A, Foster E, Brown MW, Goldenberg I, Huang DT, McNitt S, Hall WJ, Moss A, Pfeffer MA, Solomon SD; Multicenter Automatic Defibrillator Implantation Trial With Cardiac Resynchronization Therapy (MADIT-CRT) Investigators. Right ventricular function, pulmonary pressure estimation, and clinical outcomes in cardiac resynchronization therapy. Circ Heart Fail. 2013 May;6(3):435-42. doi: 10.1161/CIRCHEARTFAILURE.112.000127. Epub 2013 Mar 22. PMID 23524528

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: For this trial permission was received by several institutional review boards to include subjects death information for participants in the MADIT-CRT IDE (NCT00180271) who died between the end of the IDE and the start of the Registry. This includes 14 subjects, 7 from each arm.
Period: Overall Study
Arm/Group | MADIT-CRT ICD | MADIT-CRT CRT-D
Started | 156 | 252
Consent to Registry | 149 | 245
Completed | 144 | 237
Not Completed | 12 | 15
Not completed — Death | 11 | 12
Not completed — Withdrawal by Subject | 1 | 3

BASELINE CHARACTERISTICS:
Population: All subjects enrolled into the Reigstry were previous participants in the MADIT-CRT trial, the baseline characteristics did not pertain to the entry into the Registry.
Groups:
- Total: Total of all reporting groups
Arm/Group | MADIT-CRT ICD | MADIT-CRT CRT-D | Total
Number analyzed (Participants) | 156 | 252 | 408
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 77 | 126 | 203
  >=65 years | 79 | 126 | 205
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 78 | 114
  Male | 120 | 174 | 294
Region of Enrollment [Number; unit: participants]
  United States | 156 | 252 | 408
New York Heart Association (NYHA) Class [Number; unit: participants] — Definitions of New York Heart Association Classification:
  NYHA Class I: Asymptomatic HF: no symptoms; NYHA Class II: Mild HF: symptomatic with moderate exertion
  participants
    NYHA Class I - Ischemic | 21 | 36 | 57
    NYHA Class II - Ischemic | 54 | 87 | 141
    NYHA Class II - Non Ischemic | 81 | 129 | 210
Left Ventricular Ejection Fraction [Mean (Standard Deviation); unit: percentage] | 24 (5) | 24 (6) | 24 (6)
QRS duration [Mean (Standard Deviation); unit: milliseconds] | 158 (21) | 159 (18) | 159 (19)
Conduction disorder [Number; unit: participants]
  Left Bundle Branch Block | 110 | 181 | 291
  Right Bundle Brach Block | 22 | 31 | 53
  Nonspecific Intraventricular Conduction | 24 | 40 | 64

OUTCOME MEASURES:

1. Primary Outcome: All-Cause Mortality
Description: Outcome measured for total population. Not broken down by indication received.
Time Frame: 5 years
Measure: Number; unit: participants
Arm/Group | MADIT-CRT ICD | MADIT-CRT CRT-D
Number analyzed (Participants) | 156 | 252
participants | 11 | 12
Statistical Analysis 1: Comparison: MADIT-CRT ICD vs MADIT-CRT CRT-D; The sample size for the analysis included subjects from the original MADIT-CRT IDE (NCT00180271) that did not participate in the Registry portion, these subjects are censored at the time of study conclusion, withdrawal or death during the IDE. This was done as the Registry is a post approval continuation of the follow-up from the MADIT-CRT IDE trial. This is not a pooled analysis from separate studies; Test type: Superiority or Other; p = 0.370, Regression, Cox; Hazard Ratio (HR) = 0.88, 95% CI 2-sided [0.670 to 1.161] — The hazard ratio was calculated as the hazard rate of mortality in the CRT-D group over the hazard rate of mortality in the ICD group. A hazard ratio lower than 1 represents a reduction in relative risk of mortality for CRT-D compared to ICD
Statistical Analysis 2: Comparison: MADIT-CRT ICD vs MADIT-CRT CRT-D; These data represent the indicated sub population of left bundle branch block subjects only. (Left bundle branch block N= 110 ICD group: 181 CRT-D group); Test type: Superiority or Other; p = 0.028, Regression, Cox; Hazard Ratio (HR) = 0.68, 95% CI 2-sided [0.484 to 0.960] — The hazard ratio was calculated as the hazard rate of mortality in the CRT-D arm over the hazard rate of mortality in the ICD arm. A hazard ratio lower than 1 represents a reduction in relative risk of mortality for CRT-D compared to ICD

ADVERSE EVENTS:
Arm/Group | MADIT-CRT ICD | MADIT-CRT CRT-D
Serious Adverse Events (participants affected / at risk) | 58/149 | 93/245
Other Adverse Events (participants affected / at risk) | 9/149 | 16/245
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MADIT-CRT ICD (N=149) | MADIT-CRT CRT-D (N=245)
Laboratory Values - Abnormal (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Cancer (Blood and lymphatic system disorders) | 1 (1) | 8 (8)
Normal ERI -Device Replacement (Surgical and medical procedures) | 4 (4) | 10 (10)
Chest Pain - Ischemic (Cardiac disorders) | 0 (0) | 2 (2)
Death (General disorders) | 1 (1) | 2 (2)
Dizziness (General disorders) | 1 (2) | 2 (2)
Dyspnea (General disorders) | 4 (4) | 1 (1)
ERI - device component failure (Surgical and medical procedures) | 0 (0) | 1 (1)
Endocrine (Endocrine disorders) | 1 (1) | 1 (1)
Erosion (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Extracardiac Stimulation, Left Ventricular (Surgical and medical procedures) | 1 (1) | 1 (1)
Fatigue (General disorders) | 0 (0) | 1 (1)
Gastrointestinal (Gastrointestinal disorders) | 3 (3) | 7 (7)
Genitourinary (Renal and urinary disorders) | 7 (7) | 2 (2)
Head, Ears, Eyes, Nose and Throat (General disorders) | 0 (0) | 3 (3)
Heart Failure Symptoms (Cardiac disorders) | 23 (43) | 26 (33)
Hematological (Blood and lymphatic system disorders) | 0 (0) | 3 (3)
Hematoma (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Hypotention (Cardiac disorders) | 2 (2) | 2 (2)
Infection (> 30 days post implant procedure) (Surgical and medical procedures) | 0 (0) | 2 (2)
Integumentary (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Musculoskelatal (Musculoskeletal and connective tissue disorders) | 9 (9) | 9 (9)
Myocardial Infarction (Cardiac disorders) | 0 (0) | 4 (4)
Neurological (Nervous system disorders) | 2 (3) | 3 (3)
Lead Related, Left Ventricular (Surgical and medical procedures) | 1 (1) | 5 (5)
Patient Condition - Cardiovascular (Cardiac disorders) | 2 (2) | 2 (2)
Patient Condition - noncardiovascular (General disorders) | 2 (2) | 2 (2)
Device related, pulse generator (Surgical and medical procedures) | 2 (2) | 1 (1)
Physical Trauma (General disorders) | 0 (0) | 1 (1)
Hemorrhage, pocket (Surgical and medical procedures) | 0 (0) | 2 (2)
Pulmonary (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 4 (4)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Renal (Renal and urinary disorders) | 2 (2) | 4 (5)
Supraventricular tachycardia (Cardiac disorders) | 4 (7) | 7 (7)
Syncope (General disorders) | 1 (1) | 1 (1)
Systemic Infection (Infections and infestations) | 2 (2) | 3 (3)
Threshold Related, Left Ventricular (General disorders) | 0 (0) | 1 (1)
Thromboembolic (Vascular disorders) | 1 (1) | 7 (9)
Valvular Related (Cardiac disorders) | 0 (0) | 1 (1)
Vascular Related (Vascular disorders) | 1 (1) | 3 (3)
Ventricular Arrhythmia (Cardiac disorders) | 9 (10) | 10 (13)
Cardiogenic Shock (Cardiac disorders) | 1 (1) | 0 (0)
Hypertension (Cardiac disorders) | 1 (1) | 0 (0)
Chest Pain - Non-Cardiac (General disorders) | 4 (7) | 3 (3)
Premature Ventricular Contractions (Cardiac disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MADIT-CRT ICD (N=149) | MADIT-CRT CRT-D (N=245)
Heart Failure Symptoms (Cardiac disorders) | 9 (10) | 16 (21)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 30 days from the time submitted to the sponsor for review. The sponsor can request changes to the communication.